CLINICAL TRIAL: NCT01423981
Title: Web Based Investigation of Natural History of Keloid Disorder, an Online Survey
Status: Recruiting | Type: Observational
Sponsor: Tirgan, Michael H., M.D. (Individual)
Responsible Party: Sponsor
Other Study IDs: Tirgan 11-01
Record Dates: First submitted 2011-08-23; First posted 2011-08-26 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Keloid
Keywords: Keloid; Scar; hypertrophic scar; familial keloid
MeSH Terms: conditions — Keloid; Cicatrix; Cicatrix, Hypertrophic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with keloid disorder.: All participants have a clinical diagnosis of keloid.

SUMMARY:
This trial intends to gather very basic clinical information about keloid, its patterns of presentation, family history, ethnic background and correlation with the type of keloid, as well as prior treatment results that patients have had received.

DETAILED DESCRIPTION:
This will be a web based study, whereby patients will have to read and acknowledge the consent form online. Once patients agree and acknowledge the terms of the consent form, they will gain access to the questionnaire pages.

For those who are under age of 18, a parent or a legal guardian must sign the consent form and answer the online questions on behalf of the patient.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have clinically confirmed diagnosis of keloid
2. Adults, age over 18
3. Parent or legal guardian may participate if patient is under the age of 18
4. Able and willing to complete a web based survey

Exclusion Criteria:

* No one will be excluded from this study as long as the inclusion criteria are met.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with keloid disorder.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2011-11; Primary Completion 2030-12 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Determine the prevalence different phenotypes of keloid in participants. | Two years
  Prevalence of different phenotypes of keloid will be measured in the study population and reported. Prevalence of familial keloid in the study population will also be determined and reported. Data will be analyzed to determine the distribution of keloid among different ethic groups. Data will be analyzed to report the percentage of patients who have had one or more treatments and the percentage of patients who have had successful treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Tirgan, MD, Principal Investigator — Keloid Research Foundation
Locations (1):
- Michael H. Tirgan, MD, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All data will be shared and published

REFERENCES:
- See also: Official Study Website — http://KeloidSurvey.com